CLINICAL TRIAL: NCT06869668
Title: The Relationship Between Disability, Fear Avoidance Beliefs, Physical Performance and Quality of Life in Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Tuğba Akgüller, Principal Investigator, Istanbul Arel University
Other Study IDs: takgullereker
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Chronic Low-back Pain (cLBP)
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Correlation — Correlation between outcomes

SUMMARY:
The aim of this study was to determine the multidimensional profile of individuals with chronic low back pain (CLBP) and to determine the relationship between disability and fear avoidance beliefs, physical performance and quality of life in this population. Individuals with chronic low back pain between the ages of 18-50 will be included in the study. Disability level of the participants will be assessed with Oswestry Disability Index (ODI), fear avoidance attitudes with Avoidance Beliefs Questionnaire-Physical Activity (FABQ-PA), and quality of life with Short Form-12 (SF-12). Trunk endurance, functional mobility and static-dynamic balance will be assessed for physical performance. Trunk endurance will be assessed with McGill endurance tests, functional mobility with Timed Up and Go Test (TUG), dynamic balance with Y-balance test, and static balance with single leg stance test.

ELIGIBILITY:
Inclusion Criteria:

* Back pain for at least 3 months
* Pain intensity ≥ 3 on the Visual Analog Scale

Exclusion Criteria:

* History of spinal surgery/trauma
* Other back pain (associated with rheumatic diseases, multiple sclerosis, malignancy, etc.) instability conditions such as spondylolysis and spondylolisthesis
* Pregnancy
* Obesity (BMI ≥ 30 kg/m²)
* Presence of orthopedic problems or chronic diseases that may interfere with testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronic low back pain
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Day 1
  The questionnaire assessing the level of disability associated with low back pain includes a total of 10 questions, and each question is scored from 0 to 5. The total score ranges from 0 to 100, with higher scores indicating higher levels of disability.
Fear Avoidance Beliefs Questionnaire | Day 1
  The questionnaire, consisting of 16 items in total, has two subscales: work-related (FABQ-work) and physical activity-related (FABQ-PA). The physical activity-related subscale measures beliefs about how physical activity can affect a person's pain. The work-related subscale measures beliefs about how a person's work can affect their pain. The scale is calculated by summing the responses to all questions, with higher scores indicating higher levels of fear-avoidance beliefs.The FABQ-PA score will be used in the study.
Short Form-12/SF-12 | Day 1
  The questionnaire that evaluates the participants' health-related quality of life has two sub-scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). The PCS-12 score is obtained from the sub-dimensions of general health, physical functioning, physical role and body pain, while the PCS-12 score is obtained from the sub-dimensions of social functioning, emotional role, mental health and energy. Both the PCS-12 and PCS-12 scores range from 0 to 100, with higher scores representing better health.
McGill Trunk Muscle Endurance Tests | Day 1
  Trunk flexor endurance test: The participant is positioned by the tester with the knees and hips at 90 degrees, the trunk at 60 degrees, the hands crossed on both shoulders and the soles of the feet flat on the floor.
  Trunk extensor endurance test: Individuals are asked to hang their trunks from the bed starting from the spina iliaca anterior superior and cross both arms on the shoulders. The legs are fixed by the gastrocnemius muscle by the operator. When the individuals achieve a horizontal position, the test is started.
  Lateral Trunk Endurance Test: The individual is positioned with their feet, right arms perpendicular to the floor, elbows on the mat, left arms at chest level and left hands on the right shoulder. The test period starts as soon as they lift their hips by supporting themselves with their elbows and feet on the floor.The same is repeated for the other side.
Timed Up and Go Test (TUG) | Day 1
  A 3-meter area in front of the chair is determined. The patient is asked to get up from the chair, walk this distance, and sit down again. The elapsed time gives the result of the test and the time is recorded in seconds. The test is performed twice with a 1-minute interval and the average time is taken.
Y balance test | Day 1
  The Y balance test is a simple and reliable test used to evaluate dynamic balance. In the Y balance test, the person's balance on 3 different lines (anterior-posterolateral-posteromedial) is evaluated separately for each leg. There is a 135° angle between the anterior line and each of the posterolateral/posteromedial directions, and a 90° angle between the posterolateral and posteromedial directions. In the Y balance test, the person is positioned in the exact center of these three lines without shoes. While the foot to be tested is in the center, the other foot extends on these three different lines. The last point that can be reached without losing balance is marked each time. Three attempts are given for each direction, and the average of these three distances is recorded.
Single leg stance test | Day 1
  In the test performed for static balance assessment, the individual lifts one foot off the ground without support, with the hands on the hips. The time that the foot can be held in the air without losing balance is recorded. The test is stopped when the foot touches the ground or the hands leave the hips.
Visual Analog Scale | Day 1
  This scale is a simple and reliable scale used to record the intensity of pain felt by patients. Participants are asked to mark the level of pain they feel on the VAS, which consists of a 10 cm horizontal line extending from 0 to 10. The value of "0" on the scale indicates no pain, and the value of "10" indicates the most severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)